CLINICAL TRIAL: NCT06829160
Title: mHealth-CArdiac REhabilitation for INOCA (INOCA-CARE)
Brief Title: mHealth-CArdiac REhabilitation for INOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01040; 1R01HL170666-01 (NIH)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Ischemia
Keywords: INOCA; ANOCA; Ischemia; no obstructive coronary artery disease
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth-Cardiac Rehabilitation (CR) (Experimental): Participants in the mHealth-CR arm will receive daily therapist-directed activity and weekly phone calls, use a mHealth-CR app to track activity, heart rate and access educational materials, and use a wearable wrist activity monitoring device (such as Fitbit or Apple Watch).
  Interventions: Behavioral: Communication with exercise therapist; Behavioral: mHealth-CR; Behavioral: Wearable activity monitoring device
- Usual Care (Active Comparator): Participants in usual care arm will receive standard medical care as determined by their physician. They will also use a wearable wrist activity monitoring device.
  Interventions: Behavioral: Wearable activity monitoring device

INTERVENTIONS:
Behavioral: Communication with exercise therapist — A personalized exercise program will be designed. The assigned therapist will identify potential barriers to this plan and develop mitigation strategies. The assigned therapist will then make phone contact with participants weekly for the duration of the study. Exercise recommendations will be titrated during calls based on review of activity data.
  Arms: mHealth-Cardiac Rehabilitation (CR)
Behavioral: mHealth-CR — mHealth-CR software (currently, from Corrie Health) will permit 1) participant data entry about exercise; 2) viewing of educational material pertinent to the condition.
  Arms: mHealth-Cardiac Rehabilitation (CR)
Behavioral: Wearable activity monitoring device — Participants will be offered the Fitbit Charge 5. This commercially available product measures physical activity.

SUMMARY:
This is a multi-site phase II, 2:1 pragmatic randomized trial of 250 participants within the NYU Langone Health (NYULH) and Emory University Medical Center system to evaluate mobile health cardiac rehabilitation (mHealth-CR) in patients who meet clinical criteria for INOCA (ischemia and no obstructive coronary disease on imaging). Participants will be randomized to mHealth-CR or usual care. The study intervention takes place for 3 months which is the time period for most traditional CR programs.

The overall study goals are threefold: 1) to evaluate whether an mHealth-CR intervention that includes activity tracking, weekly counseling, and exercise documentation, improves health status (i.e., symptoms, function, and quality of life) in patients with INOCA at 3 months; 2) to evaluate effects of the mHealth-CR intervention vs. usual care on physical activity and exercise capacity, general health status, and depressive symptoms (secondary endpoints). We will also evaluate effects on primary and secondary outcomes at 6 months and 1 year; and 3) to characterize engagement and elucidate any factors that limit engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Diagnosis of Ischemia with Non-Obstructive Coronary Arteries (INOCA) based on evidence of ischemia and/or ischemic symptoms, plus non-obstructive Coronary artery disease (CAD) on computed tomography (CT) or invasive angiography

Exclusion Criteria:

* Seattle Angina Questionnaire (SAQ) = 100
* Non-ambulatory
* Pregnant
* Moderate or severe cognitive impairment
* Unable/willing to provide consent
* Incarcerated
* Unable to use mHealth
* Severe osteoarthritis or joint replacement within 3 months
* Parkinsons disease or other movement disorders
* Regular use of walker
* Life expectancy < 12 months
* Clinical judgement concerning other safety or non-adherence issues
* Unable to read and communicate in English since the app content is currently only available in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in Seattle Angina Questionnaire (SAQ) score | Baseline, Month 3
  The SAQ measures disease-related health status (functional status and quality of life) and has a four-week recall period. The SAQ generates a summary score (scale 0-100, 100 = full health, 0 = worst health).
Change in Seattle Angina Questionnaire (SAQ) score | Baseline, Month 12
  The SAQ measures disease-related health status (functional status and quality of life) and has a four-week recall period. The SAQ generates a summary score (scale 0-100, 100 = full health, 0 = worst health).
Weekly percent completion of the mHealth-CR program | Month 3
  Weekly engagement will be measured as the fraction of the following elements completed each week: exercise therapy-directed activities, daily entry of exercise data and rated perceived exertion (RPE); completed weekly phone call with exercise therapist; at least one communication with exercise therapist (outside weekly phone call); reviewing educational video/text (which will vary by week).
  Competition will be assessed as a pseudo-continuous outcome, as the score can range from 0% (0 activities completed) to 100% (all activities completed) incorporating values for each activity.

SECONDARY OUTCOMES:
Change in step count | Week 1, Month 3
  Step count is measured on a continuous basis and data will be obtained from the wearable activity monitoring device.
Change in step count | Week 1, Month 12
  Step count is measured on a continuous basis and data will be obtained from the wearable activity monitoring device.
Change in European Quality of Life Questionnaire - 5 Dimensions (EQ-5D) score | Baseline, Month 3
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Change in European Quality of Life Questionnaire - 5 Dimensions (EQ-5D) score | Baseline, Month 12
  The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Change in visual analogue scale (VAS) score | Baseline, Month 3
  VAS indicates the general health status (VAS; ranges from 0-100). Higher scores indicating the better health status.
Change in visual analogue scale (VAS) score | Baseline, Month 12
  VAS indicates the general health status (VAS; ranges from 0-100). Higher scores indicating the better health status.
Change in patient Health Questionnaire - 8 Items (PHQ-8) score | Baseline, Month 3
  The PHQ-8 is a self-reported measure of depressive symptoms composed of 8 Likert type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day), that refer to the presence of that symptom during the previous 2 weeks. The PHQ-8 final score is obtained by adding the score for each of the items, ranging from 0 to 24 (higher scores corresponding to higher levels of depression).
Change in patient Health Questionnaire - 8 Items (PHQ-8) score | Baseline, Month 12
  The PHQ-8 is a self-reported measure of depressive symptoms composed of 8 Likert type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day), that refer to the presence of that symptom during the previous 2 weeks. The PHQ-8 final score is obtained by adding the score for each of the items, ranging from 0 to 24 (higher scores corresponding to higher levels of depression).
Change in exercise time on treadmill stress test | Baseline, Month 3
  The treadmill stress test measures how well the participants heart works during physical activity. This test will take about 30 minutes in total, with about 10-15 minutes spent exercising.

OTHER OUTCOMES:
Change in rose Dyspnea Scale (RDS) score | Baseline, Month 3
  The RDS is a questionnaire that assesses how much shortness of breath a patient experiences during daily activities. The scale has four items indicating whether patients experience breathlessness with different activities (scores range from 0 to 4, with higher scores indicating dyspnea with milder activities).
Change in rose Dyspnea Scale (RDS) score | Baseline, Month 12
  The RDS is a questionnaire that assesses how much shortness of breath a patient experiences during daily activities. The scale has four items indicating whether patients experience breathlessness with different activities (scores range from 0 to 4, with higher scores indicating dyspnea with milder activities).
Change in perceived Stress Scale 4 (PSS-4) score | Baseline, Month 3
  The PSS-4 is a self-reported questionnaire consisting of four questions designed to measure how stressful a person perceives their life to be over the past month. Scores range from 0 to 16, with higher scores indicating greater perceived stress levels.
Change in perceived Stress Scale 4 (PSS-4) score | Baseline, Month 12
  The PSS-4 is a self-reported questionnaire consisting of four questions designed to measure how stressful a person perceives their life to be over the past month. Scores range from 0 to 16, with higher scores indicating greater perceived stress levels.
Number of cardiovascular hospitalizations | Month 12
  Outcome measure will be assessed through review of the electronic health record (EHR).

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: harmony.reynolds@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to harmony.reynolds@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.